CLINICAL TRIAL: NCT04599387
Title: Remote Prescribed and Monitored Exercise Program After Pulmonary Rehabilitation in Individuals With Chronic Lung Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: BIOGRADIENT LTD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-20-7416-DO-CTIL
Record Dates: First submitted 2020-10-08; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised Exercise arm (Active Comparator)
  Interventions: Other: Remote Exercise Prescription
- Usual care arm (Placebo Comparator)
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Remote Exercise Prescription — Exercise sessions will follow the recruitment meeting as prescribed by the BioGradient system, and will be tailored to the patient progress and limitations. In the beginning of each exercise session safety criteria will be collected and will allow participation . In addition, every 8 weeks and during the first exercise session outcome measurements will be collected . The study coordinator will initiate a phone call every 8 weeks to collect session data and discuss progress and limitation with the participant.
  Arms: Supervised Exercise arm
Other: Usual Care — Exercise sessions will be initiated by the patient only. In the beginning of each exercise session safety criteria will be collected and will allow participation . Every 8 weeks and once after recruitment outcome measurements will be collected . The study coordinator will initiate a phone call every 8 weeks to collect outcome session data
  Arms: Usual care arm

SUMMARY:
Remote Prescribed and Monitored Exercise Program After Pulmonary Rehabilitation in Individuals with Chronic Lung Disease

DETAILED DESCRIPTION:
The benefits of exercise during post PR (Pulmonary Rehabilitation) programs in COPD (Chronic Obstructive Pulmonary Disease) patients is well established. However, there are numerous patient's and program factors that influence the benefits gained (e.g. exercise intensity and frequency, goal setting, non-exercise modalities, compliance, social support and supervision). The investigators aim to explore the possibility of a real-life program that will allow the patient the freedom to perform exercise in their own environment. The BioGradient system allows both goal oriented, supervised exercise prescription, and the ability to adapt to the patient's schedule and preferences. The system also provides as needed human involvement for encouragement and supervision.

The investigators hypothesize that the primary outcome (the six-minute walk test, see Outcomes section) will not change significantly in active participants and measures of quality of life and adherence will be higher than reported in the literature in similar publications. Moreover, data collected may provide opportunity to explore the factors that might influence the primary and secondary outcomes, and in particular hospitalizations and exacerbations.

The current study is a patient blinded, randomized control trial, comparing usual care to goal oriented supervised post PR program. After recruitment the patient will be randomized to usual care arm or supervised exercise arm. The study duration will be 1 year (per participant), and the minimal time for each participant to be included in the final analysis will be 3 months (with at least two outcome measurements). At the end of the study each patient will be scheduled a short interview with the research coordinator for assessment of outcome measurements and spirometry testing.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for enrollment, participants must have the following inclusion criteria:

1. Age>18 years old
2. Diagnosis of COPD, based of FEV1/FVC<0.7
3. FEV1 % predicted >30%
4. Participated in PR for at least 18 sessions in the preceding year.
5. Capable of providing signed written informed consent

Exclusion Criteria:

* Participants are excluded if they have at least one of the following criteria:

  1. Currently attend (more than 5 future sessions) or eligible for a PR program
  2. On long term oxygen therapy (LTOT)
  3. Participation in another clinical study that may have an impact on the primary outcome of the current study
  4. Deemed by the healthcare team to be physically incapable of participating in the study
  5. Presence of comorbidities which, in the opinion of the healthcare team, might prevent patients from safely undertaking an exercise programme at home (for example severe orthopaedic or neurological impairments, severe cognitive impairment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in 6 Minute walk test (6MWT) | between baseline and 48weeks (end of trial)
  For this measurement the patient will be asked to performed a maximal effort for 6 minutes for which the distance walked (in meters) will be determined. To note that a self-administered 6MWT was found to yield repeatable and accurate measurement as compared to clinic administered 6MWT.

SECONDARY OUTCOMES:
Change in mean oxygen saturation | between baseline and 48weeks (end of trial)
  during 6MWT
Change in minimal oxygen saturation | between baseline and 48weeks (end of trial)
  During 6MWT
change in BORG scale | between baseline and 48weeks (end of trial)
  BORG rating of perceived exertion (RPE) at the end of the 6MWT (will be reported by a smart phone application). grade from 0 to 10, with higher numbers indicate higher perceived exertion
change in average number of steps during 6MWT | between baseline and 48weeks (end of trial)
  An average of the number of steps done per day in the preceding week before the 6MWT.
change in Modified Medical Research Council (MMRC) dyspnea scale | between baseline and 48weeks (end of trial)
  self-rating tool to measure the degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4, with higher scores indicating higher breathlessness
change in COPD Assessment Test (CAT) scale | between baseline and 48weeks (end of trial)
  measure the impact of COPD on a person's life. CAT has a scoring range of zero to 40 with higher scores indicating higher impact on person's life.
change in St. George Respiratory Questionnaire (SGRQ) | between baseline and 48weeks (end of trial)
  Disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Scores range from 0 to 100, with higher scores indicating more limitations.
Number of severe COPD exacerbation | through study completion, an average of 1 year
  Defined as any exacerbation that led to hospitalization and/or emergency department (ED) visit.
Number of moderate COPD exacerbations | through study completion, an average of 1 year
  Defined as any exacerbation treated with parenteral corticosteroids with or without antibiotics
change in FEV1/FVC | between baseline and 48weeks (end of trial)
  Will be collected during the recruitment and concluding session, and once every 6 months.
change in FVC (forced vital capacity) | between baseline and 48weeks (end of trial)
  Will be collected during the recruitment and concluding session, and once every 6 months.
change in FEV1 (forced expiratory volume in one minute) | between baseline and 48weeks (end of trial)
  Will be collected during the recruitment and concluding session, and once every 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No